CLINICAL TRIAL: NCT07188233
Title: A Study to Evaluate the Feasibility and Safety of Mitral Annular Repair With the CathHELIX™ Transcatheter System in Subjects With Functional Mitral Regurgitation
Brief Title: Mitral Annular Repair With the CathHELIX™ Transcatheter System in Subjects With FMR
Acronym: MARCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HVR Cardio Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-2023-008
Record Dates: First submitted 2025-02-28; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Mitral Valve Regurgitation (Degenerative or Functional)
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other)
  Interventions: Device: Transcatheter Mitral Valve Repair

INTERVENTIONS:
Device: Transcatheter Mitral Valve Repair — Mitral valve repair with the CathHELIX Transcatheter Mitral Annuloplasty System in subjects with functional Mitral Regurgitation

SUMMARY:
Patients with functional mitral regurgitation classified as moderate to severe (3+) or severe (4+) that are symptomatic (NYHA Class II-IV) will be evaluated for treatment using the CathHELIX Transcatheter Mitral Annuloplasty System.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe (3+) or severe (4+) functional mitral regurgitation
* Left ventricular ejection fraction ≥30%
* Symptomatic New York Heart Association (NYHA) Class II to IV).

Exclusion Criteria:

* Oxygen dependent for COPD
* Active or suspected endocarditis
* Severe symptomatic carotid stenosis
* Has undergone heart transplantation.
* Severe calcification of the mitral annulus or leaflets
* Coronary sinus anatomy that may preclude proper treatment with the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Technical Device Success (measured at the exit of the catheterization laboratory) is defined per Mitral Valve Academic Research Consortium (MVARC). | Periprocedural
  Technical Device Success: MVARC Technical Success is a definition from the Mitral Valve Academic Research Consortium for evaluating transcatheter mitral valve interventions, defined at the exit from the procedure room and requires all of the following conditions to be met:
  1. The patient is alive.
  2. There was successful access, delivery, and retrieval of the device delivery system.
  3. The first intended device was successfully deployed and correctly positioned.
  4. There was freedom from emergency surgery or reintervention related to the device or access procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Vinayak Bapat, Principal Investigator — Abbott Northwestern and United Hospitals
Locations (2):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia, Georgia
- Vilnius University Hospital, Santaros Klinikos, Public Institution, Vilnius, Lithuania, Lithuania